CLINICAL TRIAL: NCT01300364
Title: Double-blind Clinical Trial Controlled With Placebo of the Efficacy of Reboxetine and Citalopram as an Adjunct Treatment to Second Generation Antipsychotics in the Treatment of Negative Symptoms of Schizophrenia
Brief Title: Reboxetine and Citalopram as an Adjunct Treatment to Second Generation Antipsychotics in the Treatment of Negative Symptoms of Schizophrenia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundació Sant Joan de Déu (Other)
Collaborators: Centro de Investigación Biomédica en Red de Salud Mental (Network)
Responsible Party: Judith Usall Rodié, Parc Sanitari Sant Joan de Déu
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EC07/90093
Record Dates: First submitted 2011-02-18; First posted 2011-02-21 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2008-11

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Reboxetine; Citalopram; Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- sugar pill (Placebo Comparator)
  Interventions: Drug: Reboxetine; Drug: citalopram (SSRI)
- reboxetine (NRI) (Active Comparator)
  Interventions: Drug: citalopram (SSRI)
- citalopram (SSRI) (Active Comparator)
  Interventions: Drug: Reboxetine

INTERVENTIONS:
Drug: Reboxetine — 8mg/day.
  Arms: citalopram (SSRI); sugar pill
Drug: citalopram (SSRI) — 30mg/day
  Arms: reboxetine (NRI); sugar pill

SUMMARY:
Main objective: To assess the efficacy of two antidepressants of different pharmacological families: citalopram (Selective serotonin reuptake inhibitors, SSRI) and reboxetine (Norepinephrine Reuptake inhibitor, NRI) as adjunct treatments to risperidone and olanzapine for the treatment of negative symptoms of schizophrenia.

Secondary objectives: To assess the efficacy of citalopram and reboxetine as adjunct treatments to risperidone and olanzapine for the treatment of cognitive symptoms of schizophrenia. To compare the efficacy of reboxetine and citalopram as adjunct treatments for the treatment of negative and cognitive symptoms of schizophrenia.

Method: Multicentric, randomized double-blind clinical trial compared to placebo with a six months follow-up. A total of 249 patients with a diagnosis of schizophrenia (DSM-IV criteria) and significant negative symptoms, will be recruited in the 9 participating centres. Variables: sociodemographic and clinical variables (PANSS, SANS, CGI global, GAF,LSP, Hamilton scale, BACS)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia (DSM-IV criteria)
* Stable doses of antipsychotic medication (olanzapine, risperidone)for at least 60 days prior to study initiation
* Presence of significant negative symptoms (defined as one or more negative symptom score grater than 4 in the PANSS scale) (Kay 1987)
* Patients have to give written informed consent to participate in the study

Exclusion Criteria:

* Patients with a substance abuse/dependence diagnosis in the previous six months.
* Mental Retardation.
* Patients taking antidepressant in the last 4 months before the trial.
* Patients taking other antipsychotic medication, except: sinquan 100, Entumine 40, Largactil 100 and Seroquel 200.
* Patients who score more than 20 in Hamilton Rating Scale for Depression.
* Pregnancy or lactation.
* Serious impaired kidney function.
* History of hemorrhagic disorders.
* Reboxetine or citalopram allergy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Estimated)
Dates: Start 2008-11; Primary Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy end-point will be the change in the score of the PANSS negative subscale from baseline to follow-up assessment. | 24 weeks

SECONDARY OUTCOMES:
Secondary efficacy endpoints will be the change in the scores of the total PANSS and all the other clinical, social and neuropsychological scales from baseline to follow-up evaluation. | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Parc Sanitari Sant Joan de Déu, Sant Boi Llobregat, Barcelona, Spain

REFERENCES:
- [Derived] Usall J, Lopez-Carrilero R, Iniesta R, Roca M, Caballero M, Rodriguez-Jimenez R, Oliveira C, Bernardo M, Corripio I, Sindreu SD, Gonzalez Piqueras JC, Felipe AE, Fernandez de Corres B, Ibanez A, Huerta R; Abordaje Sintomas Negativos Esquizofrenia Group. Double-blind, placebo-controlled study of the efficacy of reboxetine and citalopram as adjuncts to atypical antipsychotics for negative symptoms of schizophrenia. J Clin Psychiatry. 2014 Jun;75(6):608-15. doi: 10.4088/JCP.13m08551. PMID 25004184